**Study Title:** The Effectiveness of Customised 3D-printed Insoles on Perceived Pain, Comfort, and Completion Time Among Frequent Park Runners: A Pragmatic Randomised Controlled Trial (The ZOLES Trial)

ClinicalTrials.gov identifier: NCT06034210 (https://clinicaltrials.gov/study/NCT06034210).

**Date of approval:** 04-08-2023

Consent form as approved in 'SMU\_ETHICS\_2022-23\_325' of August 4, 2023.



## **CONSENT FORM**

1.

2.

3.

4.

5.

| Name of Participant: |
|---|
| Title of the project: The effectiveness of customised 3D-printed insoles on perceived pain, comfort, and completion time among frequent Park Runners. A pragmatic randomised controlled trial (The ZOLES Trial) |
| Members of the research team: Project Lead, Sol Ibrahim 2213944@live.stmarys.ac.uk |
| Project Supervisor, Rik Mellor rik.mellor@stmarys.ac.uk Principal Investigator, Dr Filip Gertz Lysdal filip.lysdal@stmarys.ac.uk |
| I agree to take part in the above research. I have read the Participant Information Sheet which is attached to this form. I understand what my role will be in this research, and all my questions habeen answered to my satisfaction. |
| I understand that I am free to withdraw from the research at any time, for any reason and without prejudice. |
| I have been informed that the confidentiality of the information I provide will be safeguarded. |
| I am free to ask any questions at any time before and during the study. |
| I have been provided with a copy of this form and the Participant Information Sheet. |
| Data Protection: I agree to the University processing personal data which I have supplied. I agree to the processing of such data for any purposes connected with the Research Project as outlined to me. |
| Name of participant (print) |
| Signed Date |
| If you wish to withdraw from the research, please contact any investigator on the contact details |

above, or contact the trial hotline at <a href="mailto:zolesrunproject@gmail.com">zolesrunproject@gmail.com</a>